CLINICAL TRIAL: NCT06940596
Title: Exclude or Expose in Irritable Bowel Syndrome: What Works for Whom, and How? A Randomized Controlled Trial of Internet-Delivered FODMAP Diet Versus Exposure-Based Cognitive Behavioral Therapy
Brief Title: Exclude or Expose in Irritable Bowel Syndrome: What Works for Whom and How?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT31293; 2024 (Other Grant/Funding Number: Rome Foundation); APP2025943 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2025-03-31; First posted 2025-04-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome (IBS); Intestinal Diseases; Gastrointestinal Disease
Keywords: Irritable Bowel Syndrome; FODMAP Diet; Behavior Therapy; Gastrointestinal Diseases; Cognitive Behavioral Therapy; Exposure Based Cognitive Behavioral Therapy; Intestinal Diseases; Digestive System Diseases; Low FODMAP Diet
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment arms. The randomization schedule will be generated using http://www.randomization.com. Participants will be stratified by site (Australia or US) before randomization.
Who Masked: Outcomes Assessor
Masking Description: The people analyzing the results/data will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FODMAP Diet (Experimental): Fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) Diet is a 12-week online intervention with dietitian support.
  Interventions: Other: FODMAP Diet
- Exposure-based Cognitive Behavioral Therapy (E-CBT) (Experimental): Exposure-based Cognitive Behavioral Therapy is a 12-week online intervention with psychologist support.
  Interventions: Behavioral: Exposure-based Cognitive Behavioral Therapy

INTERVENTIONS:
Other: FODMAP Diet — The intervention is an online diet program. The diet is the low fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet. It is a 3-phase diet which involves: 1.Phase 1 FODMAP restriction: restrict foods high or moderate in FODMAPs and swap these for low FODMAP alternatives; 2. Phase 2 FODMAP reintroduction: continue to follow a low FODMAP diet and complete a series of food challenges to understand which foods and FODMAPs are tolerated and which trigger symptoms; 3. Phase 3 FODMAP personalization: include well-tolerated foods and FODMAPs back into the diet, and restrict poorly tolerated foods and FODMAPs to a level needed to maintain symptom relief. The online FODMAP program is a self-directed diet program with support from an online clinician (Accredited Practicing Dietitian [APD]). The content is delivered over 12 weeks. After each module participants will complete homework activities and questions and submit them to the dietitian for feedback.
  Arms: FODMAP Diet
Behavioral: Exposure-based Cognitive Behavioral Therapy — The intervention is an online behavioral therapy program. The behavioral therapy is Exposure-based Cognitive Behavioral Therapy (E-CBT) Program. The E-CBT program is organised into six steps to be completed over 12 weekly modules with support from an online clinician (Psychologist). The first step contains a rationale for the treatment and instructions on self-observation. Steps 2, 3 and 4 contain a presentation of a psychological model of IBS and continued self-observation exercises. The fifth step covers exposure exercises, divided into three categories; (1) exercises that provoke symptoms, (2) abolishment of behaviors that serve to control symptoms, (3) exposure to situations where symptoms were unwanted. The final step (Step 6) includes how to handle relapses into avoidance behaviors and how to maintain a widened behavioral repertoire. After each module participants will be directed to complete homework activities and questions and submit them to the psychologist for feedback.
  Arms: Exposure-based Cognitive Behavioral Therapy (E-CBT)

SUMMARY:
This research project will assess how two treatments for irritable bowel syndrome (one dietary and one behavioral) work and for whom. This will be done by assessing moderators (what treatment works for who and in what context) and mediators (how treatment works). Investigators will also assess how the diet and behavioral treatments affect IBS symptoms during treatment. Participants will be randomized to either: i. A FODMAP diet online program that focuses on modifying the consumption of foods high or moderate in fermentable carbohydrates (FODMAPS) to manage IBS symptoms. or, ii. An Exposure-based Cognitive Behavioral Therapy (E-CBT) online program for IBS that focuses on changing symptom-related behaviors which are known to worsen IBS symptoms.

DETAILED DESCRIPTION:
This research uses a randomized controlled trial to investigate the treatment of irritable bowel syndrome (IBS). A range of treatments for IBS are available, but each work for only a portion of patients, and it is unclear why. This research project will assess how two treatments (one dietary and one behavioral) work and for whom. Investigators will do this by assessing moderators (what treatment works for who and in what context) and mediators (how treatment works). This project will also assess how the diet and behavioral treatments affect IBS symptoms during treatment. Participants will be randomized to either: i. A FODMAP diet online program that focuses on modifying the consumption of foods high or moderate in fermentable carbohydrates (FODMAPS) to manage IBS symptoms. This treatment involves 3-phases: FODMAP restriction (phase 1), FODMAP re-introduction (phase 2), and FODMAP personalization (phase 3), or, ii. An Exposure-based Cognitive Behavioral Therapy (E-CBT) online program for IBS that focuses on symptom-related behaviors such as avoidance of activities and foods, excessive toilet visits, and behaviors to control symptoms which are known to worsen IBS symptoms. E-CBT uses daily self-observation and exposure exercises to change these behaviors to relieve IBS symptoms. Investigators believe that both treatments, FODMAP diet and E-CBT, will lead to an improvement in IBS gastrointestinal symptoms. Primary moderators and mediators to be assessed include gastrointestinal symptom anxiety, food avoidance behaviour and FODMAP intake.

ELIGIBILITY:
Inclusion Criteria: Each participant must meet all of the following criteria to be enrolled in this trial:

* Living in Australia or the United States
* Aged 18 years or older
* Body Mass Index (BMI) [Equation]18.5kg/m2 and [Equation] 34.9kg/m2
* Diagnosed with IBS by a General Practitioner, Family Physician, or Gastroenterologist, or Advanced Specialist Dietitian
* Currently fulfill Rome IV criteria for IBS
* Symptomatic at the time of recruitment (IBS-SSS > 175)
* Access to a computer and internet
* Sufficient English language and computer skills to complete a text-based online treatment
* Willing to make dietary or behavioral changes in line with the allocated treatment program
* Ability to provide informed consent

Exclusion Criteria:Patients meeting any of the following criteria will be excluded from the trial:

* Presence or known history of other GI disease (e.g. coeliac disease, Inflammatory Bowel Disease) or history of gastrointestinal cancer
* History of major gastrointestinal surgery (not appendectomy, cholecystectomy or hemorrhoidectomy)
* Individuals who report alarm symptoms (e.g., blood in stool, recent unexplained/unintentional weight loss >5% body weight, a recent change in bowel habits if >50 years, family history of gastrointestinal cancer or gastrointestinal diseases, large volumes of diarrhea occurring at night, fever associated with gut symptoms, recurrent vomiting, persistent unexplained iron deficiency) will be excluded if appropriate medical investigations have not been conducted, unless written medical approval is provided from a general practitioner, family physical, or gastroenterologist.
* Diagnosis of major disease that could explain current gastrointestinal symptoms such as severe diabetic, cardiac, liver, neurological, neuropathy disease
* History or current diagnosis of psychotic disorder or bipolar disorder
* Current diagnosis of substance abuse disorder or major depressive disorder or active suicidal ideation
* History or current diagnosis of an eating disorder
* Current enteral/parenteral feeding or use of supplemental feeds (e.g. Ensure)
* Pregnant or lactating or planning to become pregnant during the 12-week intervention period
* Commenced or change in dose of antibiotics and medications that potentially affect the gastrointestinal transit (e.g. anti-diarrheals and laxatives) in the 3 months preceding study commencement.
* Commenced taking or changed dose of probiotics, prebiotics, fibre supplements and digestive enzymes in the 3 months preceding study commencement
* Commenced or change dose in psychotropic medication in the 3 months preceding study commencement
* Are currently undertaking behavioral therapy for IBS (including cognitive behavioral therapy, CBT), or have undertaken clinician-delivered behavioral therapy for the treatment of IBS
* Are currently undertaking or have undertaken a dietitian-prescribed and delivered restrictive diet for IBS (e.g., FODMAP diet).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome (GSRS-IBS ) | Measured weekly between baseline (prior to intervention) and after intervention completed (week 12).
  The GSRS-IBS is a 13-item measure of IBS symptom severity to reflect the last 7 days. The items are scored between 1 (no discomfort at all) and 7 (very severe discomfort), rendering a total score between 13 and 91.

SECONDARY OUTCOMES:
Change from baseline in Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome (GSRS-IBS) | Baseline and 3-and 6 month follow up time points after intervention completed (week 12).
  The GSRS-IBS is a 13-item measure of IBS symptom severity to reflect the last 7 days. The items are scored between 1 (no discomfort at all) and 7 (very severe discomfort), rendering a total score between 13 and 91.
Change from baseline in Irritable Bowel Syndrome - Symptom Severity Score (IBS-SSS) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  The IBS-SSS is a 5-item measure of the severity of IBS symptoms: frequency and severity of abdominal pain, severity of bloating, dissatisfaction with bowel habits and impact on life in general. Questions ask about IBS and gut symptoms during the past 7 days except question 4 which asks participants to enter the number of days they get pain in every 10. days. A total score ranging from 0 to 500. Mild, moderate and severe cases are indicated by scores of 75 to <175, 175 to <300 and >300 respectively
Change from baseline in IBS quality of life (IBS-QOL) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  IBS-QOL is used to assess the impact on quality of life for patients with IBS and consists of 34 items scored between 1 and 5, resulting in a maximum score of 170.
Change from baseline in Nine Item ARFID (Avoidant Restrictive Food Intake Disorder) Screen (NIAS) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  NIAS is a 9-item measure of ARFID symptoms. The scale has 9 questions, scored from 0 (strongly disagree) to 5 (strongly agree) and summed into three subscales (fear of adverse consequences, lack of interest/appetite, and sensory sensitivity); each range = 0-15), with higher scores indicating greater severity.
Change from baseline in Fear of Food Questionnaire (FFQ) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  The Fear of Food Questionnaire (FFQ) is an 18-item measure of food-related fears averaged into five subscales (GI fears, food fears, food avoidance, social impairment, and distress/loss of pleasure) and a total score between 0 and 90 (each range = 0-5), with higher scores indicating greater food related fears.
Change from baseline in Patient Health Questionnaire-12 (PHQ-12) (derived from PHQ-15) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  PHQ-15 is a validated measure of somatization. Questions reflect the previous 4 weeks. It comprises 15 somatic symptoms with each symptom scored from 0 ("not bothered at all") to 2 ("bothered a lot"). The PHQ-15 will be administered to facilitate assessment of PHQ-12. The PHQ-12 is a commonly used modification of the PHQ-15 without three GI-related items; constipation, loose bowels, or diarrhea; nausea, gas, or indigestion. The PHQ-12 represents non-GI or extraintestinal somatic symptoms.
Change from baseline in Generalized anxiety disorder (GAD-7) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  GAD-7 is a 7-item questionnaire used for screening and measuring the severity of anxiety symptoms. Questions reflect the previous 14 days and responses are measured on a 4-point Likert scale; 0=not at all sure; 1=several days; 2=more than half the days; 3=nearly every day. Total GAD-7 scores range from 0-21 with higher scores indicating greater severity of symptoms.
Change from baseline in Patient Health Questionnaire (PHQ-9) questionnaire | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression severity. Questions reflect the previous 14 days. Each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day) and severity score can range from 0 to 27. PHQ-9 scores of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline in Gastrointestinal Specific Anxiety (GSA) measured using Visceral Sensitivity Index (VSI) | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  The VSI is a 15-item measure of gastrointestinal-specific anxiety, scored on a Likert scale of 1 to 6 with 1=strongly agree; 2=moderately agree; 3=mildly agree; 4=mildly disagree; 5=moderately disagree and 6=strongly disagree.
Change from baseline in Avoidance behavior measured using Irritable Bowel Syndrome-Behavioural Responses Questionnaire (IBS-BRQ) | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  IBS-BRQ is a 26-item measure of avoidance behavior. The scale has 26 items, scored from 1 (never) to 7 (always), indicating how persistently the particular avoidance or toilet behavior is carried out.
Change from baseline in Total FODMAP intake measured using 3-day food diary | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  Participants will record their food intake for 3 days (including one weekend day) using paper or an app. Total FODMAP intake will be calculated g/day.
Change from baseline in stool frequency and consistency using 7-day stool diary based on Bristol Stool Form Scale (BSFS) | Baseline, after intervention completed (week 12), and at follow up time points of 3-and 6 months following the 12-week intervention.
  The stool diary will be completed over 7 days and is based on the Bristol Stool Form Scale (BSFS) for IBS subtyping and bowel habit assessment i.e. stool frequency and consistency. Stool consistency will be quantified according to ROME classifications.
Gastrointestinal microbiome composition and function using stool sample using OMNIgene GUT | Gastrointestinal microbiome composition and function will be measured 2nd weekly between baseline (prior to intervention) and after intervention completed (week 12) as exploratory mediators.
  Gut microbiome composition (i.e., alpha diversity, beta diversity, relative abundance) and function 16S rRNA and shotgun sequencing. Measured as exploratory mediators.
Individual FODMAPs' intake using 3-day food diary | Will be measured 2nd weekly between baseline (prior to intervention) and after intervention completed (week 12) as exploratory mediators.
  Participants will record their food intake for 3 days (including one weekend day) using paper or an app. Individual FODMAPs' intake will be calculated g/day. Measured as exploratory mediators.
Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome GSRS-IBS | Baseline (prior to start of intervention) as an exploratory moderator.
  The GSRS-IBS is a 13-item measure of IBS symptom severity to reflect the last 7 days. The items are scored between 1 (no discomfort at all) and 7 (very severe discomfort), rendering a total score between 13 and 91. Measured as an exploratory moderator.
IBS quality of life (IBS-QOL) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  Description: I IBS-QOL is used to assess the impact on quality of life for patients with IBS and consists of 34 items scored between 1 and 5, resulting in a maximum score of 170. Measured as an exploratory moderator.
Fear of Food Questionnaire (FFQ) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  The Fear of Food Questionnaire (FFQ) is an 18-item measure of food-related fears averaged into five subscales (GI fears, food fears, food avoidance, social impairment, and distress/loss of pleasure) and a total score between 0 and 90 (each range = 0-5), with higher scores indicating greater food related fears. Measured as an exploratory moderator.
Nine Item ARFID (Avoidant Restrictive Food Intake Disorder) Screen (NIAS) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  NIAS is a 9-item measure of ARFID symptoms. The scale has 9 questions, scored from 0 (strongly disagree) to 5 (strongly agree) and summed into three subscales (fear of adverse consequences, lack of interest/appetite, and sensory sensitivity); each range = 0-15), with higher scores indicating greater severity. Measured as an exploratory moderator.
Patient Health Questionnaire-12 (PHQ-12) (derived from PHQ-15) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  PHQ-15 is a validated measure of somatization. Questions reflect the previous 4 weeks. It comprises 15 somatic symptoms with each symptom scored from 0 ("not bothered at all") to 2 ("bothered a lot"). The PHQ-15 will be administered to facilitate assessment of PHQ-12. The PHQ-12 is a commonly used modification of the PHQ-15 without three GI-related items; constipation, loose bowels, or diarrhea; nausea, gas, or indigestion. The PHQ-12 represents non-GI or extraintestinal somatic symptoms. Measured as an exploratory moderator.
Patient Health Questionnaire (PHQ-9) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression severity. Questions reflect the previous 14 days. Each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day) and severity score can range from 0 to 27. PHQ-9 scores of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depression, respectively. Measured as an exploratory moderator.
Generalized anxiety disorder (GAD-7) questionnaire | Baseline (prior to start of intervention) as an exploratory moderator.
  GAD-7 is a 7-item questionnaire used for screening and measuring the severity of anxiety symptoms. Questions reflect the previous 14 days and responses are measured on a 4-point Likert scale; 0=not at all sure; 1=several days; 2=more than half the days; 3=nearly every day. Total GAD-7 scores range from 0-21 with higher scores indicating greater severity of symptoms. Measured as an exploratory moderator.
Gastrointestinal microbiome composition and function using stool sample using a stool sample collection kit. | Baseline (prior to start of intervention) as an exploratory moderator.
  Gut microbiome composition (i.e., alpha diversity, beta diversity, relative abundance) and function 16S rRNA and shotgun sequencing . Measured as an exploratory moderator.
IBS subtype using 7-day stool diary based on Bristol Stool Form Scale (BSFS). | Baseline (prior to start of intervention) as an exploratory moderator.
  The stool diary will be completed over 7 days and is based on the Bristol Stool Form Scale (BSFS) for IBS subtyping and bowel habit assessment i.e. stool frequency and consistency. Stool consistency will be quantified according to ROME classifications. Measured as a exploratory moderator.
Client Satisfaction Questionnaire | End of the 12-week intervention and at 3-and 6 months follow up time points after 12-week intervention..
  The Client Satisfaction Questionnaire is an 8-question brief global measure of client satisfaction. The eight questions are measured on a 4-point Likert scale with questions 1, 3, 6 and 7 measured on a positive scale and questions 2, 4, 5 and 8 on a negative scale. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Proportion of participants who achieve a change from baseline in Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome (GSRS-IBS) of >30% total score | Baseline and after intervention completed (week 12)
  The GSRS-IBS is a 13-item measure of IBS symptom severity to reflect the last 7 days. The items are scored between 1 (no discomfort at all) and 7 (very severe discomfort), rendering a total score between 13 and 91.
Proportion of participants who achieve a change from baseline in Irritable Bowel Syndrome - Symptom Severity Score (IBS-SSS) of ≥50 points total score. | Baseline and after intervention completed (week 12)
  The IBS-SSS is a 5-item measure of the severity of IBS symptoms: frequency and severity of abdominal pain, severity of bloating, dissatisfaction with bowel habits and impact on life in general. Questions ask about IBS and gut symptoms during the past 7 days with the exception of question 4 which asks participants to enter the number of days they get pain in every 10. days. A total score ranging from 0 to 500. Mild, moderate and severe cases are indicated by scores of 75 to <175, 175 to <300 and >300 respectively

OTHER OUTCOMES:
Gastrointestinal Specific Anxiety (GSA) measured using Visceral Sensitivity Index (VSI) | VSI will be measured 2nd weekly between baseline (prior to intervention), after intervention (week 12) and and at follow up timepoints of 3-and 6 months following the 12-week intervention as a putative mediator.
  The VSI is a 15-item measure of gastrointestinal-specific anxiety, scored on a Likert scale of 1 to 6 with 1=strongly agree; 2=moderately agree; 3=mildly agree; 4=mildly disagree; 5=moderately disagree and 6=strongly disagree. The VSI is being measured as a putative mediator.
Avoidance behavior measured using Irritable Bowel Syndrome-Behavioural Responses Questionnaire (IBS-BRQ) | IBS-BRQ will be measured 2nd weekly between baseline (prior to intervention), after intervention (week 12) and and at follow up timepoints of 3-and 6 months following the 12-week intervention as a putative mediator.
  IBS-BRQ is a 26-item measure of avoidance behavior. The scale has 26 items, scored from 1 (never) to 7 (always), indicating how persistently the particular avoidance or toilet behavior is carried out. IBS-BRQ is measured as a putative mediator.
Total FODMAP intake measured using 3-day food diary | Total FODMAP intake will be measured 2nd weekly between baseline (prior to intervention), after intervention (week 12) and and at follow up timepoints of 3-and 6 months following the 12-week intervention as a putative mediator.
  Participants will record their food intake for 3 days (including one weekend day) using paper or an app. Total FODMAP intake will be calculated g/day. Total FODMAP intake is being measured as a putative mediator.
Treatment preference | Baseline (prior to start of intervention) as a putative moderator.
  Baseline treatment preference will be assessed with a single question prior to randomization: "If you had a choice, which treatment would you prefer to receive?". Three response options will be provided: FODMAP diet program; Cognitive Behavioral Therapy program; No preference. Measured as a putative moderator.
Gastrointestinal Specific Anxiety (GSA) measured using Visceral Sensitivity Index (VSI) | Baseline (prior to start of intervention) as a putative moderator.
  The VSI is a 15-item measure of gastrointestinal-specific anxiety, scored on a Likert scale of 1 to 6 with 1=strongly agree; 2=moderately agree; 3=mildly agree; 4=mildly disagree; 5=moderately disagree and 6=strongly disagree. The VSI is being measured as a putative moderator.
Avoidance behavior measured using Irritable Bowel Syndrome-Behavioural Responses Questionnaire (IBS-BRQ) | Baseline (prior to start of intervention) as a putative moderator.
  IBS-BRQ is a 26-item measure of avoidance behavior. The scale has 26 items, scored from 1 (never) to 7 (always), indicating how persistently the particular avoidance or toilet behavior is carried out. IBS-BRQ is measured as a putative moderator.
Total FODMAP intake measured using 3-day food diary | Baseline (prior to start of intervention) as a putative moderator.
  Participants will record their food intake for 3 days (including one weekend day) using paper or an app. Total FODMAP intake will be calculated g/day. Total FODMAP intake is being measured as a putative mediator. Measured as a putative moderator.
Credibility expectancy questionnaire (CEQ) questionnaire | End of week 2 of 12-week intervention
  The Credibility & Expectancy Questionnaire is a 6-question measure of treatment expectancy and credibility. Credibility is derived from the first three 'think' (cognitively based) questions and expectancy is derived from the fourth 'think' question and the two 'feel' (affectively based) questions. Measured as a control variable.
Working alliance inventory for guided internet intervention (WAI-I) questionnaire | End of week 2 of 12-week intervention
  The Working Alliance Inventory for guided Internet interventions (WAI-I) is a 12 item tool to evaluate the working alliance in the context of guided Internet interventions. It consists of two subscale dimensions; Dimension 1: task and goal agreement with the program; and Dimension 2: bond with therapist. Items are rated on a 5-point Likert scale ranging from 1 (never) to 5 (always) and will be reported as a total score. Measured as a control variable.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Jessica Biesiekierski, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Potential data shared includes:
  * Individual participant data that underlie the results reported in the article after de-identification (text, tables, figures and appendices)
  * Trial protocol
  * Statistical Analysis Plan
  * Participant Information Consent Form
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available beginning 3 months following analysis and article publication for 15 years.
Access Criteria: The IPD and supporting information will be made available for use by future researchers from a recognized research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept University of Melbourne conditions for access.
URL: https://figshare.unimelb.edu.au/

REFERENCES:
- [Background] Biesiekierski JR, Manning LP, Murray HB, Vlaeyen JWS, Ljotsson B, Van Oudenhove L. Review article: exclude or expose? The paradox of conceptually opposite treatments for irritable bowel syndrome. Aliment Pharmacol Ther. 2022 Aug;56(4):592-605. doi: 10.1111/apt.17111. Epub 2022 Jul 1. PMID 35775328